CLINICAL TRIAL: NCT04126148
Title: Breathing-Maneuver-Induced Myocardial Oxygenation Reserve Validated by FFR (B-MORE)
Acronym: B-MORE
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Matthias Friedrich, Cardiologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2019-4137
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Stenosis
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Age matched Healthy participants (150): Healthy Participants Age: > 40y No known current or pre-existing significant medical problems that would affect the cardiovascular or respiratory system
- Coronary Artery Disease (CAD) Patients (200): Coronary Artery Disease (CAD) Patients Age > 18 y Patients with an Indication for invasive coronary angiography based on symptoms and a test positive for inducible coronary ischemia, or previous coronary angiography.

SUMMARY:
The study aims to determine a diagnostic marker for regionally impaired myocardial oxygenation response in patients with suspected coronary artery stenosis.

DETAILED DESCRIPTION:
This observational applied research international study aims to assess the validity of breathing maneuvers as a vasoactive maneuver and Oxygenation-Sensitive Cardiac Magnetic Resonance Imaging (OS-CMR) in a patient population. OS-CMR results will be compared to the clinical gold standard of Fractional Flow Reserve (FFR) and instant wave-free ratio (iFR) as a secondary objective, to determine if this non-invasive, no pharmaceutical agent imaging technique can identify areas of oxygenation deficit in myocardium perfused by a stenosed coronary artery.

ELIGIBILITY:
Inclusion Criteria:

Healthy Participants

* Age: > 40y
* No known current or pre-existing significant medical problems that would affect the cardiovascular or respiratory system.

CAD Patients

* Age > 18 y
* Indication for invasive coronary angiography based on symptoms and a test positive for inducible coronary ischemia, or previous coronary angiography.

Exclusion Criteria:

ALL participants:

* General MRI contraindications: Pacemakers, defibrillating wires, implanted defibrillators, intracranial aneurysm clips, metallic foreign bodies in the eyes, knowledge or suspicion of pregnancy.
* Consumption of caffeine (coffee, tea, cocoa, chocolate, "energy drink") during the 12 hours prior to the exam.
* Regular nicotine consumption during the last 6 months.

Patients only

* Vasoactive medication (e.g. nitro) during the 12 hours prior to the exam Contraindications to adenosine (2nd or 3rd A-V block, sinus node disease, asthma, bronchoconstrictive diseases).
* Acute Coronary Syndrome (ACS), or previous Coronary Artery Bypass Surgery
* Previous myocardial infarction within 1 month
* Clinically unstable condition
* Significant or uncontrolled arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be composed of patients with suspected or known CAD and healthy volunteers. The primary group will consist of patients with 1- or 2-vessel CAD. Patients diagnosed with 3-vessel or no obstructive disease in an angiography visit after the CMR exam will be included as a sub-group, with not more than 25% of the study population being in this group. Healthy volunteers will serve to act as a control for the assessment of a diagnostic cut-off.
  Patient who performed the CMR and then the angiography, who are deemed to have no obstructive (no vessel) CAD or 3-vessel CAD, will be assigned to a subgroup of the study. No vessel disease will be those who have no vessel stenosis of >0.75. 3-vessel disease will be those who have a stenosis of >0.75 in all three coronary arteries.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
B-MORE: Diagnostic cut-off - Relative change of myocardial signal intensity | 2019-2022
  To obtain a diagnostic cut-off of the mean Breathing-Maneuver-induced Myocardial Oxygenation REserve (B-MORE) of a coronary territory as defined by the relative change of myocardial signal intensity (delta SI[%]) in oxygenation-sensitive CMR (OS-CMR) images, at the 15s and 30s time point of a post-hyperventilation breath-hold for detecting an associated severe coronary artery stenosis as defined by FFR of less than 0.75 or a QCA assessment of >0.75, as compared to the global delta SI[%] in age-matched healthy volunteers

SECONDARY OUTCOMES:
30sec B-MORE Cut-off | 2019-2022
  A student's t-test will assess a cut-off of the Breathing maneuver induced Myocardial Oxygenation REserve (MORE), at the 30s time point of the breath hold, for a region perfused by a stenosed coronary artery (FFR / iFR or QCA >0.75) as compared to a healthy coronary artery (FFR / iFR or QCA <0.75), within a patient.
Heart rate response to hyperventilation. | 2019-2022
  Markers of diagnostic accuracy will be obtained to assess the accuracy the heart rate response to hyperventilation.
Myocardial strain response at the 15s and 30s time point during breath-hold | 2019-2022
  Markers of diagnostic accuracy will be obtained to assess the accuracy of the myocardial strain response at the 15s and 30s time point of the breath-hold
Accuracy of B-MORE and strain response at the 15s and 30s time point of the breath-hold | 2019-2022
  Markers of diagnostic accuracy will be obtained to assess the accuracy of a combination of the B-MORE and the strain response at the 15s and 30s time point of the breath-hold
B-MORE - strain response at 15s and 30s time breath hold and Heart rate response | 2019-2022
  Markers of diagnostic accuracy will be obtained to assess the accuracy of a combination of the B-MORE, the strain response at the 15s and 30s time point of the breath-hold, and the heart rate response to hyperventilation
Relationship between B-MORE vs heart rate response to hyperventilation | 2019-2022
  A student's t-test will assess the relationship between B-MORE results and heart rate response to hyperventilation
Relationship between myocardial strain and Heart rate | 2019-2022
  A student's t-test will assess the relationship between the strain response at the 15 and 30 s timepoints and heart rate response to hyperventilation
Relationship between B-MORE and myocardial strain measurements -each coronary territory | 2019-2022
  A student's t-test will assess the relationship between B-MORE results and myocardial strain measurements (circumferential, longitudinal, and radial) at the 15s and 30s time point for each coronary territory.
Global relationship between B-MORE results and myocardial strain measurements | 2019-2022
  A student's t-test will assess the global relationship between B-MORE results and myocardial strain measurements (circumferential, longitudinal, and radial).
Relationship between B-MORE and QCA | 2019-2022
  Pearson's correlation coefficient will be obtained to assess the relationship between B-MORE results at the 15s and 30s time point of the breath-hold and Quantitative Coronary Angiography (QCA) measurements for each coronary territory.
Relationship between B-MORE and FFR / iFR | 2019-2022
  Pearson's correlation coefficient will be obtained to assess the relationship between B-MORE results at the 15 s and 30s time point of the breath-hold and FFR / iFR measurements for each coronary territory.
Relationship between B-MORE (15s and 30s) vs QCA | 2019-2022
  Pearson's correlation coefficient will be obtained to assess the relationship between B-MORE results after hyperventilation and Quantitative Coronary Angiography (QCA) measurements for each coronary territory.
Relationship between B-MORE vs FFR - iFR each coronary territory | 2019-2022
  To assess the relationship between B-MORE results after hyperventilation and FFR / iFR measurements for each coronary territory.
Relationship between B-MORE vs T1/T2 mapping | 2019-2022
  Pearson's assess the relationship between B-MORE results and global T1/T2 mapping measurements.
Breathing maneuver - Clinical feasibility | 2019-2022
  Recorded time, exclusion rate due to inability to perform the breathing maneuvers, will be reported for clinical feasibility during MRI and while performing iFR. Any serious adverse effects of the breathing maneuver will be reported for safety.
B-MORE analysis intra and inter-reader reproducibility | 2019-2022
  Correlation coefficients will be obtained to evaluate the intra- and inter-reader reproducibility of B-MORE.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias G Friedrich, MD, Principal Investigator — Reseach Institute of the McGill University health Center
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided